CLINICAL TRIAL: NCT00494338
Title: A Phase II Trial of Docetaxel and Celecoxib in Patients With Androgen Independent Prostate Cancer
Brief Title: Phase II Trial of Docetaxel and Celecoxib in Patients With Androgen Independent Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to celecoxib safety issues
Sponsor: Sanofi (Industry)
Responsible Party: Study medical Officer, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976J_2504
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic Androgen Independent Prostate Cancer (MAIPC)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: Docetaxel

SUMMARY:
A multi-center controlled, non-comparative open Phase II trial of docetaxel and celecoxib in patients with metastatic androgen independent prostate cancer where efficacy is measured by PSA response defined as a 50% reduction in PSA maintained on two consecutive evaluations at least 4 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed MAIPC
* Documented progressive disease in bone, soft tissue or PSA despite castrate levels of testosterone
* If LHRH agonist were used previously it must be kept
* Previous anti-androgen should be held at least 4 weeks for flutamida or cyproterone and 6 weeks for bycalumida
* Previous DES should be held for at least 4 weeks before partcipating in the trial
* Chemotherapy naive patients
* No prior radioisotope
* Less than 25% of bone marrow should be irradiated for prior palliative radiotherapy
* KPS> 70%
* Adequate hematologic, hepatic and renal function

Exclusion Criteria:

* Patients with serious medical illness
* History of significant active cardiac disease
* History of gastrointestinal ulceration, bleeding or perforation
* History of myocardial infarctin within past 12 months
* Allergy to sulfonamides or to celecoxib or history of urticaria to any NSAID

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-11; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of docetaxel and celecoxib by PSA response defined as a 50% reduction in PSA maintained on two consecutive evaluations at least 4 weeks apart | two consecutive evaluations at least 4 weeks apart

SECONDARY OUTCOMES:
Response in measurable disease by response evaluation criteria in solid tumors (RECIST) criteria, time to progression, overall survival and toxicity by Natonal Cancer Institute Commum Toxicity Criteria version 2.0. | response evaluation criteria in solid tumors (RECIST) criteria, time to progression, overall survival and toxicity by Natonal Cancer Institute Commum Toxicity Criteria version 2.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, M.D., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, São Paulo, Brazil